CLINICAL TRIAL: NCT05448365
Title: The Use of Vitamin D in Combination With Epigallocatechin Gallate, D-chiro-inositol and Vitamin B6 in the Treatment of Women With Uterine Fibroid
Brief Title: Vitamin D, Epigallocatechin Gallate, D-chiro-inositol and Vitamin B6 in Uterine Fibroid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DELPHYS PLUS
Record Dates: First submitted 2022-07-04; First posted 2022-07-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Uterine Fibroids; D-chiro-inositol; Inositol; Epigallocatechin Gallate; Vitamin D; Vitamin B6
MeSH Terms: conditions — Leiomyoma | interventions — epigallocatechin gallate; Vitamin D; Vitamin B 6

STUDY DESIGN:
Intervention Model Description: Women with uterine fibroids
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be a double-clind, placebp-controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGCG, Vit D, DCI, Vit B6 (Active Comparator): Women with uterine fibroids randomized to treatment group
  Interventions: Dietary Supplement: Epigallocatechin gallate, Vitamin D, Vitamin B6, D-chiro-inositol
- Placebo (Placebo Comparator): Women with uterine fibroids randomized to placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Epigallocatechin gallate, Vitamin D, Vitamin B6, D-chiro-inositol — The patients will take for three months two tablets per day each containing 150mg epigallocatechin gallate, 25 mg D-chiro-inositol, 5mg Vitamin B6 and 25μg Vitamin D
  Arms: EGCG, Vit D, DCI, Vit B6
Dietary Supplement: Placebo — Maltodextrines
  Arms: Placebo

SUMMARY:
The study will evaluate the impact on uterine fibroids' volume of a combination of natural molecules including Epigallocatechin gallate, Vitamin D, D-chiro-inositol and Vitamin B6.

The patients will be evaluated at baseline and after three months of treatment with placebo or product.

ELIGIBILITY:
Inclusion Criteria:

1. uterine fibroid with diameter greater than or equal to 4cm or multiple fibroids
2. eligible for surgery
3. symptoms like menometrorrhagia or pelvic pain

Exclusion Criteria:

1. BMI>30
2. currently pregnant or breastfeeding
3. diabetic
4. suspect of malignancy
5. diagnosis of cancer

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Diameter | 3 months
  Greater diameter of the diagnosed uterine fibroids

SECONDARY OUTCOMES:
Volume | 3 months
  Total volume of the diagnosed uterine fibroids
Need for surgery | 3 months
  The percentage of patients that decide to avoid surgery
pVEGF-R | 3 months
  the phosphorilation of VEGF receptor
Marker of cellular proliferation | 3 months
  expression of ki67, ER, PR

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale Dario camberlingo, Francavilla Fontana, Apulia
  - Ospedale Veris Delli Ponti, Scorrano, Apulia

IPD SHARING:
Plan to Share IPD: No